CLINICAL TRIAL: NCT06009016
Title: Inflammation and Coagulation Factors in Cerebrospinal Fluid for Predicting Persistent Cerebral Edema After Subarachnoid Hemorrhage
Brief Title: Inflammation and Coagulation Factors for Predicting Cerebral Edema After SAH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Yuanjian Fang, Second Affiliated Hospital, School of Medicine, Zhejiang University, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2023-059
Record Dates: First submitted 2023-08-13; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Inflammation; Coagulation and Hemorrhagic Disorders; Cerebral Edema
MeSH Terms: conditions — Inflammation; Thrombosis; Hemorrhagic Disorders; Brain Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Inflammatory factors and coagulation factors level in cerebrospinal fluid after subarachnoid hemorrhage — Inflammatory factors and coagulation factors level in cerebrospinal fluid will be tested by ELISA kits.

SUMMARY:
Explore the role of Inflammation and coagulation factors in cerebrospinal fluid for predicting persistent cerebral edema after subarachnoid hemorrhage

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage patients admitted to our neurosurgery department with modified Fisher Scale 3-4, with a confirmed radiographic diagnosis.

Exclusion Criteria:

* Angiogram-negative patients, patients with a history of trauma or previous brain injury (stroke, hemorrhage, surgery et al. which left associated chronic changes on CT), arteriovenous malformation, radiological data lost, accompany with serious comorbidities before subarachnoid hemorrhage onset (such as coagulation defects, uncontrollable hypertension, and arrhythmia et.al.), initial radiological data performed more than 3 days after SAH onset

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subarachnoid hemorrhage patients admitted to our neurosurgery department with modified Fisher Scale 3-4, with a confirmed radiographic diagnosis. Age range from 20-80.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral edema after subarachnoid hemorrhage | At 3 and 7days after SAH onset
  Cerebral edema after subarachnoid hemorrhage will be determined by the SEBES score. SEBES 0-2 is mild edema; SEBES 3-4 is severe edema.
Outcome at 3 months after subarachnoid hemorrhage | 3 months after subarachnoid hemorrhage
  Outcome will be determined by the modified Rankin Score (mRS). mRS 0-2 is favorable outcome; mRS3-5 is poor outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided